CLINICAL TRIAL: NCT04872621
Title: Calquence 100 mg Capsules General Drug Use-Results Study; All Patient Investigation in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia (Including Small Lymphocytic Lymphoma)
Brief Title: Calquence CLL rr Japan PMS_Japan Post-Marketing Surveillance (PMS) Study - All Patient Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8224C00001
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia (Including Small Lymphocytic Lymphoma)
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To understand the incidence of ADRs of Calquence 100 mg capsules (acalabrutinib) used in patients with relapsed or refractory chronic lymphocytic leukaemia (including small lymphocytic lymphoma) in a real-world post-marketing setting

DETAILED DESCRIPTION:
To understand the incidence of ADRs of Calquence 100 mg capsules (acalabrutinib) used in patients with relapsed or refractory chronic lymphocytic leukaemia (including small lymphocytic lymphoma) in a real-world post-marketing setting.

This investigation will be conducted for application for re-examination specified in Article 14-4 of the Pharmaceutical Affairs Law. In addition, after launch, the data for a certain number of all cases are collected and the survey is required to be conducted for all cases as conditions of approval.

ELIGIBILITY:
Inclusion Criteria:

Patients with relapsed or refractory chronic lymphocytic leukemia (small lymphocytic lymphoma) who are treated with the product -

Exclusion Criteria:

None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsed or refractory chronic lymphocytic leukaemia (small lymphocytic lymphoma) who are treated with the product
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs | 52weeks
  the incidence of ADRs related to Calquence Safety specifications: Haemorrhage, infection, bone narrow depression, arrhythmia, ischemic heart disease, tumour lysis syndrome, interstitial lung disease, and second primary malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (40):
- Japan (40):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluatedas per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes,indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level datain an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8224C00001&attachmentIdentifier=c4a80b38-f15c-4a88-8cbe-e94a6b7f8078&fileName=Clinical_Study_Report_(CSR)_Synopsis,_RIMS_CAL_D8224C00001.pdf&versionIdentifier=